CLINICAL TRIAL: NCT05663554
Title: Improving Glycemic Control Using a Virtual Weight Control Program Among Adults With Type 2 Diabetes
Acronym: VITAL-2
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study sponsor cancelled funding prior to enrolment due to competing priorities.
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: WW International Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #PBRC 2022-048
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WW Intervention (Experimental): Participants in the intervention arm will be contacted by a WW Coach and will receive a voucher code that provides 12 months of access to the WW program and instructions for redeeming the code. The program will include access to weekly Virtual Workshops and the WW App. WW is a widely available, commercial behavioral weight management program that encourages healthy habits in the areas of food, activity, mindset, and sleep, with topics specific to diabetes.
  Interventions: Behavioral: WW Intervention
- Usual Care (Active Comparator): Patients in the Usual Care Arm will continue to receive routine medical care by their healthcare provider. In addition, at the baseline visit, participants in the Usual Care Arm will receive one 50-minute virtual on-line session of nutrition counseling with a registered dietitian, with additional materials at the time of their 6- and 12-month follow-up assessments, based on current recommendations of the American Diabetes Association
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: WW Intervention — The core of the WW food program is the SmartPoints® system. Briefly, the SmartPoints® system assigns each food and beverage a SmartPoints® value per volume based on four components: calories, sugar, saturated fat, and protein. Certain foods have a SmartPoints® value of zero (ZeroPoint foods). These foods (e.g., lean sources of protein such as skinless chicken breast and vegetables) form the basis of a healthy eating pattern, are at low risk for overconsumption and do not have to be weighed, measured or tracked. Participants were assigned a personalized SmartPoints® Budget, based on reported food and lifestyle preferences, and designed to create an energy deficit, using the Mifflin St-Jeor formula, which uses age, sex, height, and weight to estimate resting energy expenditure.
  Arms: WW Intervention
Other: Usual Care — The Usual Care group will continue to receive routine medical care by their provider, in addition to receiving one 50-minute virtual on-line session of nutrition counseling with a registered dietitian, with additional materials at the time of their 6- and 12-month follow-up assessments.
  Arms: Usual Care

SUMMARY:
The study is a randomized clinical trial with the primary aim of determining the effectiveness of the WW intervention at reducing HbA1c in patients with type 2 diabetes.

DETAILED DESCRIPTION:
This study is a 12-month, two-arm, parallel controlled trial. Up to 486 adults with overweight or obesity and type 2 diabetes will be randomized to either 1) intervention or 2) usual care. The intervention arm will participate in a WW program which will include access to weekly Virtual Workshops and the WW App. WW is a widely available, commercial behavioral weight management program that encourages healthy habits in the areas of food, activity, mindset, and sleep, with topics specific to diabetes. Participants in the usual care arm will receive their normal, usual care from their healthcare providers in addition to a session with a Registered Dietician at baseline. All patients will participate in the collection of patient-reported outcomes at baseline and at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 18.0 - 74.9 years of age
* Participant-reported diagnosis of type 2 diabetes
* HbA1c 7.0%-11% (inclusive)
* Overweight or obesity (BMI 25-50 kg/m2)
* On stable regimen of medications that can affect weight or diabetes outcomes for at least 3 months (brief regimens of medications such as antibiotics, steroids, etc. are permitted)
* Willingness to attend weekly WW Virtual Workshops and participate in WW Digital program
* Access to a smartphone/tablet that can download the WW app
* Willing and able to provide a valid email address for use in the study
* Be able to communicate (oral and written) in English
* Be under the care of a physician who will be responsible for managing the subject's diabetes and a participant who is willing to give release to provide their treating MD with information about the trial
* Be able to provide informed consent

Exclusion Criteria:

* Participation in a weight control program within the past 3 months
* Weight loss of ≥ 5 kg in the previous 6 months
* Taking prescription or over-the-counter weight loss medications within last 3 months
* History of weight loss surgery
* History of major surgery within three months of enrollment
* Type 1 diabetes
* Renal insufficiency consisting of potassium over 5.5 mmol/L on a non-hemolyzed specimen, or a creatinine > 2.5 mg/dL
* Albumin < 3 g/dL
* Alanine Aminotransferase > 3 times the upper limit of normal (normal range is 7-56 IU/L)
* More than 1 severe hypoglycemic event (requiring emergency medical services) in the past 12 months, unless the participant's physician provides written clearance for participation
* Hemoglobinopathy that interferes with measurement of HbA1c
* Class II or higher congestive heart failure
* Unstable heart disease (an ongoing workup or treatment for a cardiac symptom such as unstable angina, coronary ischemia)
* Presence of implanted cardiac defibrillator
* Blood pressure ≥160/100 mm Hg. If a potential participant has a blood pressure ≥160/100 mm Hg it is acceptable to re-test this potential participant within one week of the original test
* Thyroid disease for which the participant is untreated or has had treatment changed within the last 6 months. History of thyroid disease or current thyroid disease treated with a stable medication regimen for at least 2 months is acceptable
* Orthopedic limitations that would interfere with ability to engage in regular physical activity
* Uncontrolled gastrointestinal disorders including chronic malabsorptive conditions, peptic ulcer disease, Crohn's disease, chronic diarrhea or active gallbladder disease
* Current cancer or cancer treatment, or a history of cancer or cancer treatment within the last 3 years. Persons with successfully resected non-melanoma carcinoma of the skin may be enrolled
* Dementia, psychiatric illness, or substance abuse that may interfere with adherence (e.g., illness that is currently unstable or resistant to first-line therapy; substance abuse in the past year)
* History of clinically diagnosed eating disorder including anorexia nervosa or bulimia nervosa.
* Women who are pregnant, lactating, trying to become pregnant or unwilling to use an effective means of birth control
* Currently consuming >14 alcoholic drinks (1 drink = 12 fl oz beer, 4 fl oz wine or 1.5 fl oz liquor) per week and unwilling to limit intake to less than 3 drinks per day during study participation
* Participation in another clinical trial within 30 days prior to enrollment
* Participation in WW anytime since November 2021
* Any other condition or factor which in the opinion of the study physician or investigator makes it inadvisable for the candidate to participate in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c% at 6 months | Baseline and 6 months.
  Hemoglobin A1c levels (%) are measured using standard laboratory methods
Change in HbA1c% at 12 months | Baseline and 12 months.
  Hemoglobin A1c levels (%) are measured using standard laboratory methods

SECONDARY OUTCOMES:
Percent weight loss at 6 months | Baseline and 6 months
  Body weight is measured using standard methods with the patient wearing light clothing
Percent weight loss at 12 months | Baseline and 12 months
  Body weight is measured using standard methods with the patient wearing light clothing
Change in waist circumference at 6 months | Baseline and 6 months
  Waist circumference is measured using standard methods with an inelastic tape
Change in waist circumference at 12 months | Baseline and 12 months
  Waist circumference is measured using standard methods with an inelastic tape
Change in systolic blood pressure at 6 months | Baseline and 6 months
  Systolic blood pressure is measured using standard clinical methods
Change in systolic blood pressure at 12 months | Baseline and 12 months
  Systolic blood pressure is measured using standard clinical methods
Change in diastolic blood pressure at 6 months | Baseline and 6 months
  Diastolic blood pressure is measured using standard clinical methods
Change in diastolic blood pressure at 12 months | Baseline and 12 months
  Diastolic blood pressure is measured using standard clinical methods
Change in total cholesterol at 6 months | Baseline and 6 months
  Total cholesterol is assayed using standard laboratory methods
Change in total cholesterol at 12 months | Baseline and 12 months
  Total cholesterol is assayed using standard laboratory methods
Change in high-density lipoprotein cholesterol at 6 months | Baseline and 6 months
  High-density lipoprotein cholesterol is assayed using standard laboratory methods
Change in high-density lipoprotein cholesterol at 12 months | Baseline and 12 months
  High-density lipoprotein cholesterol is assayed using standard laboratory methods
Change in low-density lipoprotein cholesterol at 6 months | Baseline and 6 months
  Low-density lipoprotein cholesterol is estimated using standard laboratory methods
Change in low-density lipoprotein cholesterol at 12 months | Baseline and 12 months
  Low-density lipoprotein cholesterol is estimated using standard laboratory methods
Change in triglycerides at 6 months | Baseline and 6 months
  Triglycerides are assayed using standard laboratory methods
Change in triglycerides at 12 months | Baseline and 12 months
  Triglycerides are assayed using standard laboratory methods
Change in physical activity at 6 months | Baseline and 6 months
  Physical activity is assessed with the Global Physical Activity Questionnaire. A valid and reliable instrument from the World Health Organization that measures physical activity intensity, duration, and frequency in three domains: occupational physical activity, transport-related physical activity, and physical activity during discretionary or leisure time. It also captures sedentary time. There are 16 questions.
Change in physical activity at 12 months | Baseline and 12 months
  Physical activity is assessed with the Global Physical Activity Questionnaire. A valid and reliable instrument from the World Health Organization that measures physical activity intensity, duration, and frequency in three domains: occupational physical activity, transport-related physical activity, and physical activity during discretionary or leisure time. It also captures sedentary time. There are 16 questions.
Change in dietary intake at 6 months | Baseline and 6 months
  Dietary Intake will be assessed using DietID (www.DietID.com). DietID harnesses diet quality photo navigation technology to identify participant's dietary intake by showing a series of images that participants select based on what reflects their current dietary pattern. Once a pattern is identified, DietID provides nutrient intake data and a Healthy Eating Index 2015 score.
Change in dietary intake at 12 months | Baseline and 12 months
  Dietary Intake will be assessed using DietID (www.DietID.com). DietID harnesses diet quality photo navigation technology to identify participant's dietary intake by showing a series of images that participants select based on what reflects their current dietary pattern. Once a pattern is identified, DietID provides nutrient intake data and a Healthy Eating Index 2015 score.
Change in perceived stress at 6 months | Baseline and 6 months
  Perceived stress is measured using the Perceived Stress Scale, a 10-item questionnaire that measures the extent to which a participant's life is unpredictable, uncontrollable, and overloading. It was designed for use in older adolescents and adults, and is considered to have adequate internal reliability and construct validity. Each question asks about how the participant has felt or thought in the past month and uses a 5-point Likert scale (0=never, 4=very often). Scores are calculated by summing responses and higher scores indicate greater perceived stress.
Change in perceived stress at 12 months | Baseline and 12 months
  Perceived stress is measured using the Perceived Stress Scale, a 10-item questionnaire that measures the extent to which a participant's life is unpredictable, uncontrollable, and overloading. It was designed for use in older adolescents and adults, and is considered to have adequate internal reliability and construct validity. Each question asks about how the participant has felt or thought in the past month and uses a 5-point Likert scale (0=never, 4=very often). Scores are calculated by summing responses and higher scores indicate greater perceived stress.
Change in diabetes distress at 6 months | Baseline and 6 months
  The Diabetes Distress Scale contains 17 total items with 4 subscales: Emotional Burden (items 1, 3, 8, 11, 14), Physician-related distress (items 2, 4, 9, 15), Regimen-related distress (items 5, 6, 10, 12, 16), and Interpersonal distress (7, 13, 17). The total score is calculated by taking an average of participant responses to all 17 items. In the same manner, each subscale can have its own score by taking an average of subscale specific participant responses. A mean item score of 3 or higher is considered moderate distress and a level of distress worthy of clinical attention. The Diabetes Distress scale has been tested for reliability and validity in US based populations and abroad.
Change in diabetes distress at 12 months | Baseline and 12 months
  The Diabetes Distress Scale contains 17 total items with 4 subscales: Emotional Burden (items 1, 3, 8, 11, 14), Physician-related distress (items 2, 4, 9, 15), Regimen-related distress (items 5, 6, 10, 12, 16), and Interpersonal distress (7, 13, 17). The total score is calculated by taking an average of participant responses to all 17 items. In the same manner, each subscale can have its own score by taking an average of subscale specific participant responses. A mean item score of 3 or higher is considered moderate distress and a level of distress worthy of clinical attention. The Diabetes Distress scale has been tested for reliability and validity in US based populations and abroad.
Change in quality of life at 6 months | Baseline and 6 months
  The Impact of Weight on Quality of Life-Lite is a validated self-report measure for an individual's perception of how their weight affects their day-to-day life. Respondents rate the degree to which their weight affects them on 31 items using a five-point Likert scale (1, never true; 2, rarely true; 3, sometimes true; 4, usually true; 5, always true). The IWQOL-Lite consists of 5 scales (physical function, self-esteem, sexual life, public distress, and work).
Change in quality of life at 12 months | Baseline and 12 months
  The Impact of Weight on Quality of Life-Lite is a validated self-report measure for an individual's perception of how their weight affects their day-to-day life. Respondents rate the degree to which their weight affects them on 31 items using a five-point Likert scale (1, never true; 2, rarely true; 3, sometimes true; 4, usually true; 5, always true). The IWQOL-Lite consists of 5 scales (physical function, self-esteem, sexual life, public distress, and work).
Change in well-being at 6 months | Baseline and 6 months
  Well-being will be measured using the World Health Organization-5 Well-being Index, which consists of five statements, which respondents rate, in relation to the past two weeks, using a six-point Likert scale (0, at no time; 1, some of the time; 2, less than half of the time; 3, more than half of the time; 4, most of the time; 5, all of the time). The total raw score ranges from 0 to 25, and is multiplied by 4 to give the final score, with 0 representing the worse imaginable well-being and 100 representing the best imaginable well-being.
Change in well-being at 12 months | Baseline and 12 months
  Well-being will be measured using the World Health Organization-5 Well-being Index, which consists of five statements, which respondents rate, in relation to the past two weeks, using a six-point Likert scale (0, at no time; 1, some of the time; 2, less than half of the time; 3, more than half of the time; 4, most of the time; 5, all of the time). The total raw score ranges from 0 to 25, and is multiplied by 4 to give the final score, with 0 representing the worse imaginable well-being and 100 representing the best imaginable well-being.
Change in habit strength at 6 months | Baseline and 6 months
  Habit strength will be assessed with the Self-Report Behavioral Automaticity Index, a 4-item measure that that is reliable, correlates highly with existing measures, and is sensitive to effects that characterize habits. The 4-items assess whether Behavior X is something... "I do automatically", "I do without having to consciously remember", "I do without thinking", and "I start doing before I realize I'm doing it". Items are scored using a 7-point Likert scale ranging from strongly disagree to strongly agree.
Change in habit strength at 12 months | Baseline and 12 months
  Habit strength will be assessed with the Self-Report Behavioral Automaticity Index, a 4-item measure that that is reliable, correlates highly with existing measures, and is sensitive to effects that characterize habits. The 4-items assess whether Behavior X is something... "I do automatically", "I do without having to consciously remember", "I do without thinking", and "I start doing before I realize I'm doing it". Items are scored using a 7-point Likert scale ranging from strongly disagree to strongly agree.
Change in emotional eating at 6 months | Baseline and 6 months
  Emotional eating will be measured with the Palatable Eating Motives Scale- Coping Subscale, which measures intentionally using palatable food to cope with negative feelings and has demonstrated reliability, convergent validity and discriminant validity. The coping subscale additionally demonstrated incremental validity with BMI. The coping subscale consists of 4 questions with response options Almost Never/Never to Almost always/Always.
Change in emotional eating at 12 months | Baseline and 12 months
  Emotional eating will be measured with the Palatable Eating Motives Scale- Coping Subscale, which measures intentionally using palatable food to cope with negative feelings and has demonstrated reliability, convergent validity and discriminant validity. The coping subscale additionally demonstrated incremental validity with BMI. The coping subscale consists of 4 questions with response options Almost Never/Never to Almost always/Always.
Change in hunger at 6 months | Baseline and 6 months
  Hunger will be measured using the Hunger Visual Analogue Scale, which is a reliable measure for appetite research. The Hunger Visual Analogue Scale asks "How hungry did you feel over the past week" and is composed of a line with words anchored at each end describing the extremes (Not at all hungry, Extremely hungry). Participants are asked to make a mark on the line corresponding to their feelings and quantification of the measurement is done by measuring the distance from the left end of the mark.
Change in hunger at 12 months | Baseline and 12 months
  Hunger will be measured using the Hunger Visual Analogue Scale, which is a reliable measure for appetite research. The Hunger Visual Analogue Scale asks "How hungry did you feel over the past week" and is composed of a line with words anchored at each end describing the extremes (Not at all hungry, Extremely hungry). Participants are asked to make a mark on the line corresponding to their feelings and quantification of the measurement is done by measuring the distance from the left end of the mark.
Change in diabetes medications at 6 months | Baseline and 6 months
  The number of diabetes medications is summed at each time point
Change in diabetes medications at 12 months | Baseline and 12 months
  The number of diabetes medications is summed at each time point
Change in proportion of patents achieving an HbA1c% <=6.5% at 6 months | Baseline and 6 months
  Hemoglobin A1c levels (%) are measured using standard laboratory methods
Change in proportion of patents achieving an HbA1c% <=6.5% at 12 months | Baseline and 12 months
  Hemoglobin A1c levels (%) are measured using standard laboratory methods
Change in proportion of patents achieving an HbA1c% <=7% at 6 months | Baseline and 6 months
  Hemoglobin A1c levels (%) are measured using standard laboratory methods
Change in proportion of patents achieving an HbA1c% <=7% at 12 months | Baseline and 12 months
  Hemoglobin A1c levels (%) are measured using standard laboratory methods
Change in food cravings at 6 months | Baseline and 6 months
  Food cravings will be assessed using the Food Cravings Inventory, a 33-item self-report measure designed to assess the subjective experience of food craving across 33 different foods. The measure consists of 5 empirically-derived factors: high fats, sweets, carbohydrates, starches, fast food fats, & fruits and vegetables. The questionnaire is scaled in a frequency format, assessing the frequency with which an individual experiences a craving for a particular food. All items are scored in the following manner: Never = 1, Rarely = 2, Sometimes = 3, Often = 4, & Always=5. Fat = Average of items 3,4,7,11,17,23,31,32. Sweet=Average of items 1,9,15,19,20,27,28,30. Carb=Average of items 6,10,14,16,22,25,26,33. FFF=Average of items 2,8,13,24. FCI-Fr/Veg=Average of items 5,12,18,21,29. Total=Average of all 33 items.
Change in food cravings at 12 months | Baseline and 12 months
  Food cravings will be assessed using the Food Cravings Inventory, a 33-item self-report measure designed to assess the subjective experience of food craving across 33 different foods. The measure consists of 5 empirically-derived factors: high fats, sweets, carbohydrates, starches, fast food fats, & fruits and vegetables. The questionnaire is scaled in a frequency format, assessing the frequency with which an individual experiences a craving for a particular food. All items are scored in the following manner: Never = 1, Rarely = 2, Sometimes = 3, Often = 4, & Always=5. Fat = Average of items 3,4,7,11,17,23,31,32. Sweet=Average of items 1,9,15,19,20,27,28,30. Carb=Average of items 6,10,14,16,22,25,26,33. FFF=Average of items 2,8,13,24. FCI-Fr/Veg=Average of items 5,12,18,21,29. Total=Average of all 33 items.
Change in self compassion at 6 months | Baseline and 6 months
  Self-compassion will be assessed using the Self-Compassion Scale, a 26-item measure of self-compassion that is psychometrically valid and theoretically coherent. The scale consists of six subscales: self-kindness, self-judgement, common humanity, isolation, mindfulness, and over-identified. Subscales are computed by calculating the mean of subscale item responses. A total self-compassion score can be obtained by reverse scoring the negative subscale items (self-judgement, isolation, and over-identification) and computing a grand mean of all six subscale means.
Change in self compassion at 12 months | Baseline and 12 months
  Self-compassion will be assessed using the Self-Compassion Scale, a 26-item measure of self-compassion that is psychometrically valid and theoretically coherent. The scale consists of six subscales: self-kindness, self-judgement, common humanity, isolation, mindfulness, and over-identified. Subscales are computed by calculating the mean of subscale item responses. A total self-compassion score can be obtained by reverse scoring the negative subscale items (self-judgement, isolation, and over-identification) and computing a grand mean of all six subscale means.
Change in restraint/disinhibition at 6 months | Baseline and 6 months
  The Three Factor Eating Questionnaire- Restraint and Disinhibition subscales measures cognitive restraint of eating and disinhibition. The scales contain 37 items and have been tested for reliability and validity. Higher scores indicate greater levels of restraint or disinhibition.
Change in restraint/disinhibition at 12 months | Baseline and 12 months
  The Three Factor Eating Questionnaire- Restraint and Disinhibition subscales measures cognitive restraint of eating and disinhibition. The scales contain 37 items and have been tested for reliability and validity. Higher scores indicate greater levels of restraint or disinhibition.
Change in body appreciation at 6 months | Baseline and 6 months
  The Body Appreciation Scale measures individuals acceptance of, favorable opinions toward, and respect for their bodies. The scale demonstrates internal consistency, convergent validity, incremental validity, and discriminant validity. Measurement invariance upheld across sexes and US sample types (college vs. community samples). There are 10 items, each assessed on a scale from 1-never to 5-always.
Change in body appreciation at 12 months | Baseline and 12 months
  The Body Appreciation Scale measures individuals acceptance of, favorable opinions toward, and respect for their bodies. The scale demonstrates internal consistency, convergent validity, incremental validity, and discriminant validity. Measurement invariance upheld across sexes and US sample types (college vs. community samples). There are 10 items, each assessed on a scale from 1-never to 5-always.
Change in weight bias at 6 months | Baseline and 6 months
  The Weight Bias Internalization Scale has 13 items and responses are rated on a 7-point Likert scale (strongly disagree -strongly agree). Responses provide insight on the participant's internalized beliefs and feelings regarding their weight. There are two subscales: Weight-Related Distress (7 items; 7-13; Cronbach's alpha =0.910) and Weight-Related Self-Devaluation (6 items; 1-6; Cronbach's alpha =0.763). The scale has been tested for validity in people with overweight and obesity and the two factor model demonstrated good to excellent fit with the data. Scores are calculated by taking an average of the response values. Questions 1,2,4,5, should be reverse scored before calculating the average.
Change in weight bias at 12 months | Baseline and 12 months
  The Weight Bias Internalization Scale has 13 items and responses are rated on a 7-point Likert scale (strongly disagree -strongly agree). Responses provide insight on the participant's internalized beliefs and feelings regarding their weight. There are two subscales: Weight-Related Distress (7 items; 7-13; Cronbach's alpha =0.910) and Weight-Related Self-Devaluation (6 items; 1-6; Cronbach's alpha =0.763). The scale has been tested for validity in people with overweight and obesity and the two factor model demonstrated good to excellent fit with the data. Scores are calculated by taking an average of the response values. Questions 1,2,4,5, should be reverse scored before calculating the average.

CONTACTS AND LOCATIONS:
Overall Officials: Peter T Katzmarzyk, PhD, Principal Investigator — Pennington Biomedical Research Center; Monica L Baskin, PhD, Principal Investigator — University of Pittsburgh Health Sciences; Jamy D Ard, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (3):
- United States (3):
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Wake Forest University Health Sciences, Greensboro, North Carolina
  - University of Pittsburgh Health Sciences, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
A de-identified individual-level dataset will be made available to researchers making a reasonable request to the principal investigator. Data will be made available 1 year after publication of the primary outcomes manuscript.
Supporting Information: Study Protocol
Time Frame: Data and supporting information will be available 1 year after the publication of the primary outcome paper.
Access Criteria: Upon reasonable request to the Principal Investigator.